CLINICAL TRIAL: NCT05644353
Title: A Bioequivalence Study of Subcutaneous Injections of Mirikizumab Reference Solution Using Investigational 1-mL and 2-mL Prefilled Syringes and Mirikizumab Test Solution Formulation Using Investigational 1-mL and 2-mL Prefilled Syringes in Healthy Participants
Brief Title: A Bioequivalence Study of Mirikizumab (LY3074828) Solution in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17773; I6T-MC-AMBY (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab (Experimental): Participants received 3 milliliter (mL) mirikizumab as 2 subcutaneous (SC) injections of 1 mL and 2 mL delivered via Pre-filled Syringe (PFS) to abdomen or arms or thighs on Day 1.
  Interventions: Drug: Mirikizumab
- Citrate-Free Mirikizumab (Experimental): Participants received 3 mL citrate- free mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to abdomen or arms or thighs on Day 1.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered SC.
  Other Names: LY3074828

SUMMARY:
The main purpose of this study is to evaluate amount of mirikizumab (test) that gets into the blood stream and how long it takes the body to get rid of it, when given via pre-filled syringe compared to mirikizumab (reference) solution given via pre-filled syringe. The information about any adverse effects experienced will be collected and the tolerability of mirikizumab will also be evaluated.

Screening is required within 35 days prior to enrolment. For each participant, the total duration of the clinical trial will be about 17 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Have a body mass index( BMI) within the range of 18.0 to 34.0 kg/m2, inclusive.
* Are males or non-pregnant women of childbearing potential (WOCBP) or women not of childbearing potential (WNOCBP).

Exclusion Criteria:

* Have significant allergies to humanized monoclonal antibodies or known allergies to mirikizumab, related compounds or any components of the formulation, or history of significant atopy
* Have an abnormal blood pressure, pulse rate, or temperature as determined by the investigator
* Intend to use over-the-counter or prescription medication, including herbal medications and traditional medications, within 7 days prior to dosing
* Are lactating or pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Qps-Mra, Llc, Miami, Florida
  - Axis, Dilworth, Minnesota
  - Labcorp Clinical Research LP, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otani Y, Feagan BG, D'Haens GR, Escobar R, Morris NJ, Payne CD, Ugolini Lopes M, Zhang X. Pharmacokinetic Comparability and Safety Between Original and Citrate-Free Mirikizumab Formulations for Subcutaneous Injections: Results from Three Clinical Trials. Adv Ther. 2025 May;42(5):2369-2384. doi: 10.1007/s12325-025-03158-y. Epub 2025 Mar 21. PMID 40117091

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirikizumab - Abdomen: Participants received 3 milliliter (mL) mirikizumab as 2 subcutaneous (SC) injections of 1 mL and 2 mL delivered via Pre-filled Syringe (PFS) in the abdomen on Day 1.
- Mirikizumab - Arm: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to arms on Day 1.
- Mirikizumab - Thigh: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to thighs on Day 1.
- Citrate-Free Mirikizumab - Abdomen: Participants received 3 mL citrate-free mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to the abdomen on Day 1.
- Citrate-Free Mirikizumab - Arm: Participants received 3 mL citrate-free mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to arms on Day 1.
- Citrate-Free Mirikizumab - Thigh: Participants received 3 mL citrate-free mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to thighs on Day 1.
Period: Overall Study
Arm/Group | Mirikizumab - Abdomen | Mirikizumab - Arm | Mirikizumab - Thigh | Citrate-Free Mirikizumab - Abdomen | Citrate-Free Mirikizumab - Arm | Citrate-Free Mirikizumab - Thigh
Started | 74 | 76 | 76 | 75 | 75 | 74
Received At Least One Dose of Study Drug | 74 | 76 | 76 | 75 | 75 | 74
Completed | 72 | 74 | 75 | 75 | 74 | 74
Not Completed | 2 | 2 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Mirikizumab - Abdomen: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS in the abdomen on Day 1.
- Total: Total of all reporting groups
Arm/Group | Mirikizumab - Abdomen | Mirikizumab - Arm | Mirikizumab - Thigh | Citrate-Free Mirikizumab - Abdomen | Citrate-Free Mirikizumab - Arm | Citrate-Free Mirikizumab - Thigh | Total
Number analyzed (Participants) | 74 | 76 | 76 | 75 | 75 | 74 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.9) | 41.9 (13.4) | 41.5 (11.9) | 40.3 (12.5) | 41.4 (12.5) | 40.8 (12.5) | 40.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 50 | 41 | 36 | 38 | 35 | 238
  Male | 36 | 26 | 35 | 39 | 37 | 39 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 48 | 48 | 45 | 44 | 44 | 271
  Not Hispanic or Latino | 32 | 27 | 28 | 30 | 31 | 30 | 178
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 2 | 4
  Asian | 2 | 1 | 0 | 0 | 3 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 8 | 12 | 9 | 12 | 13 | 67
  White | 56 | 62 | 62 | 64 | 56 | 53 | 353
  More than one race | 2 | 1 | 1 | 0 | 1 | 1 | 6
  Unknown or Not Reported | 1 | 2 | 1 | 2 | 3 | 1 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 76 | 76 | 75 | 75 | 74 | 450

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab in a Citrate-free Solution Formulation Compared to the Solution Formulation
Description: PK: Cmax of Mirikizumab
Time Frame: Pre-dose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704 and, 2040 hours post day 1 dose
Population: All participants who received at least one dose of study drug and had evaluable PK data for this outcome. Per protocol, PK analysis was performed to compare all mirikizumab participants together versus all citrate-free mirikizumab participants together.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- Mirikizumab: Participants received 3 mL mirikizumab as 2 SC injections of 1 mL and 2 mL delivered via PFS to abdomen or arms or thighs on Day 1.
Arm/Group | Mirikizumab | Citrate-Free Mirikizumab
Number analyzed (Participants) | 207 | 208
micrograms per milliliter (μg/mL) | 20.9 (43) | 20.9 (39)

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Mirikizumab in a Citrate-free Solution Formulation Compared to the Solution Formulation
Description: PK: AUC[0-∞] of Mirikizumab
Time Frame: Pre-dose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704 and, 2040 hours post day 1 dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/ mL
Arm/Group | Mirikizumab | Citrate-Free Mirikizumab
Number analyzed (Participants) | 205 | 208
microgram*day per milliliter (μg*day/ mL | 331 (39) | 325 (36)

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Mirikizumab in a Citrate-free Solution Formulation Compared to the Solution Formulation
Description: PK: AUC[0-tlast] of Mirikizumab
Time Frame: Pre-dose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704 and, 2040 hours post day 1 dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/ mL
Arm/Group | Mirikizumab | Citrate-Free Mirikizumab
Number analyzed (Participants) | 205 | 208
microgram*day per milliliter (μg*day/ mL | 327 (39) | 320 (36)

ADVERSE EVENTS:
Time Frame: Baseline Through Follow-Up (Up To 13 Weeks)
Description: All participants who have received at least one dose of study drug.
Arm/Group | Mirikizumab - Abdomen | Mirikizumab - Arm | Mirikizumab - Thigh | Citrate-Free Mirikizumab - Abdomen | Citrate-Free Mirikizumab - Arm | Citrate-Free Mirikizumab - Thigh
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76 | 0/76 | 0/75 | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76 | 0/76 | 0/75 | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 27/74 | 38/76 | 36/76 | 11/75 | 17/75 | 17/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirikizumab - Abdomen (N=74) | Mirikizumab - Arm (N=76) | Mirikizumab - Thigh (N=76) | Citrate-Free Mirikizumab - Abdomen (N=75) | Citrate-Free Mirikizumab - Arm (N=75) | Citrate-Free Mirikizumab - Thigh (N=74)
Injection site reaction (General disorders) | 19 (30) | 31 (57) | 31 (56) | 6 (10) | 12 (20) | 12 (21)
Medication error (Injury, poisoning and procedural complications) | 6 (12) | 6 (12) | 5 (10) | 5 (10) | 5 (10) | 4 (8)
Headache (Nervous system disorders) | 3 (7) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05644353/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT05644353/SAP_001.pdf